CLINICAL TRIAL: NCT05795244
Title: A Phase II Study of Induction PD-1 Blockade (Nivolumab) in Patients With Surgically Complete Resectable Mismatch Repair Deficient Endometrial Cancer (NIVEC)
Brief Title: Study of Induction PD-1 Blockade (Nivolumab) in Patients With Surgically Complete Resectable Mismatch Repair Deficient Endometrial Cancer (NIVEC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, JUNGYUN LEE, M.D, PhD, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-0001
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Endometrial Neoplasms; Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — - Nivolumab 480 mg/every 4 weeks/IV infusion/6 cycles
  Other Names: Opdivo

SUMMARY:
phase 2 clinical trial to confirm the pathological complete response rate of PD-1 blocker use in patients with Mismatch Repair Deficiency(MMRd) endometrial cancer that can be completely resected surgically.

DETAILED DESCRIPTION:
Multi-center, non-randomized, open-label, A Phase II study of induction PD-1 blockade (nivolumab) in patients with surgically completely resectable mismatch repair deficient endometrial cancer. A total of 30 subjects from 7 institutions in Korea will be enrolled in this trial.

Patients will be administered Nivolumab 480mg intravenously every 4 weeks for a total 6 cycles. After the 6 cycles of anti-cancer therapy, surgical resection will be performed. If clinical and pathological complete response is confirmed, it is possible to observe the patient's progress without surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Explicit and voluntary consent to participation in the trial obtained by signing and dating a consent form that clearly and completely describes the purpose, potential risks, and other important issues related to the trial.
2. Sex: female
3. Age (at the time of informed consent): 20 years and older
4. Subjects with histologically-or cytologically-confirmed endometrial cancer or carcinosarcoma(Mixed Mullerian Tumor)
5. Clinical stage: Stage I - IIIC2 and surgically completely resectable
6. No evidence of distant metastases
7. MMRd or MSI-H subtype (defined by either deficient/loss expression of mismatch repair (MMR) proteins MLH1, PMS2, MSH2, MSH6 or microsatellite instability-high (MSI-H) by polymerase chain reaction assay for 5 microsatellite markers)
8. ECOG Performance Status Score 0 or 1
9. Patients with a life expectancy of at least 3 months
10. Patients whose latest laboratory data meet the below criteria within 7 days before first dose. If the date of the laboratory tests at the time of enrollment is not within 7 days before the first dose of the investigational product, testing must be repeated within 7 days before the first dose of the investigational product, and these latest laboratory tests must meet the following criteria. Of note, laboratory data will not be valid if the patient has received a granulocyte colony-stimulating factor (G CSF) or blood transfusion within 14 days before testing.

    * White blood cells ≥2,000/mm3 and neutrophils ≥1,500/mm3
    * Platelets ≥100,000/mm3
    * Hemoglobin ≥9.0 g/dL
    * AST (GOT) and ALT (GPT) ≤3.0-fold the upper limit of normal (ULN) of the study site (or ≤5.0-fold the ULN of the study site in patients with liver metastases)
    * Total bilirubin ≤1.5-fold the ULN of the study site
    * Creatinine ≤1.5-fold the ULN of the study site or creatinine clearance (either the measured or estimated value using the Cockcroft-Gault equation) >45 mL/min
11. Women of childbearing potential (including women with chemical menopause or no menstruation for other medical reasons)#1 must agree to use contraception#2 from the time of informed consent until 5months or more after the last dose of the investigational product. Also, women must agree not to breastfeed from the time of informed consent until 5 months or more after the last dose of the investigational product.

    * Women of childbearing potential are defined as all women after the onset of menstruation who are not postmenopausal and have not been surgically sterilized (e.g., hysterectomy, bilateral tubal ligation, bilateral oophorectomy). Post-menopause is defined as amenorrhea for ≥12 consecutive months without specific reasons. Women using oral contraceptives, intrauterine devices, or mechanical contraception such as contraceptive barriers are regarded as having childbearing potential.
    * The subject must consent to use any one of the following methods of contraception: a condom for the subject's partner (male), an intrauterine device (IUD) for female subjects, or skin implantation of a rod contraceptive (Implanon).
    * Complete sexual abstinence is also acceptable: Sexual abstinence is considered highly effective only if it is defined as abstaining from sexual intercourse with the opposite sex for the entire duration of the trial treatment-related risks. The reliability of sexual abstinence in relation to the duration of the trial needs to be evaluated, and sexual abstinence should be a preferred and routine lifestyle of the subjects.

Exclusion Criteria:

1. Patients with multiple primary cancers (with the exception of completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, or superficial bladder cancer, or any other cancer that has not recurred for at least 5 years)
2. Patients with residual adverse effects of prior therapy or effects of surgery that would affect the safety evaluation of the investigational product in the opinion of the investigator or sub-investigator.
3. Patients with current or past history of severe hypersensitivity to any other antibody products
4. Patients with concurrent autoimmune disease or history of chronic or recurrent autoimmune disease
5. Patients with a current or past history of interstitial lung disease or pulmonary fibrosis diagnosed based on imaging or clinical findings. Patients with radiation pneumonitis may be randomized if the radiation pneumonitis has been confirmed as stable (beyond acute phase) without any concerns about recurrence.
6. Patients with concurrent diverticulitis or symptomatic gastrointestinal ulcerative disease
7. Patients with pericardial fluid, pleural effusion, or ascites requiring treatment
8. Patients with uncontrollable, tumor-related pain
9. Patients who have experienced a transient ischemic attack, cerebrovascular accident, thrombosis, or thromboembolism (pulmonary arterial embolism or deep vein thrombosis) within 180 days before randomization
10. Patients with a history of uncontrollable or significant cardiovascular disease meeting any of the following criteria:

    * Myocardial infarction within 180 days before randomization
    * Uncontrollable angina pectoris within 180 days before randomization
    * New York Heart Association (NYHA) Class III or IV congestive heart failure
    * Uncontrollable hypertension despite appropriate treatment (e.g., systolic blood pressure ≥150mmHg or diastolic blood pressure ≥ 90 mmHg lasting 24 hours or more)
    * Arrhythmia requiring treatment
11. Patients receiving or requiring anticoagulant therapy for a disease. Patients receiving antiplatelet therapy including low-dose aspirin may be enrolled.
12. Patients with uncontrollable diabetes mellitus
13. Patients with systemic infections requiring treatment
14. Patients who have received systemic corticosteroids (except for temporary use, e.g., for examination or prophylaxis of allergic reactions) or immunosuppressants within 28 days before randomization
15. Patients who have received antineoplastic drugs (e.g., chemotherapy agents, molecular-targeted therapy agents, or immunotherapy agents) within 28 days before randomization
16. Patients who have undergone surgical adhesion of the pleura or pericardium within 28 days before randomization
17. Patients who have undergone surgery under general anesthesia within 28 days before randomization
18. Patients who have undergone surgery involving local or topical anesthesia within 14 days before randomization
19. Patients who have received radiotherapy within 28 days before randomization, or radiotherapy to bone metastases within 14 days before randomization
20. Patients who have received any radiopharmaceuticals (except for examination or diagnostic use of radiopharmaceuticals) within 56 days before randomization
21. Patients with a positive test result for any of the following: HIV-1 antibody, HIV-2 antibody, HTLV-1 antibody, HBs antigen, or HCV antibody
22. Patients with a negative HBs antigen test but a positive test result for either HBs antibody or HBc antibody with a detectable level of HBV-DNA
23. Women who are pregnant or breastfeeding, or possibly pregnant
24. Patients who have received any other unapproved drug (e.g., investigational use of drugs, unapproved combined formulations, or unapproved dosage forms) within 28 days before randomization
25. Patients who have previously received Nivolumab, anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD L2 antibody, anti-CD137 antibody, anti-CTLA-4 antibody or other therapeutic antibodies or pharmacotherapies for regulation of T-cells
26. Patients judged to be incapable of providing consent for reasons such as concurrent dementia
27. Other patients judged by the investigator or sub-investigator to be inappropriate as subjects of this study
28. Patient with current or past history of hypersensitivity to Nivolumab.
29. WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response | At 3 months
  Tumor response evaluation will be conducted based on imaging tests and pathological response of the endometrium. The evaluation of endometrium should be performed using Dilatation & Currettage or hysteroscopic biopsy every 3 cycles.

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 3 months
  Objective response rate is defined according to RECIST v1.1 or iRECIST.
Progression free survival (PFS) | 1 year
  PFS is defined as the time from treatment start until the first documented sign of disease progression or death from any cause.
Overall survival (OS) | Approximately up to 6 years.
  OS is defined as the time from first treatment until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: JUNGYUN LEE, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee YJ, Lee YY, Park JY, Cho HW, Lim MC, Kim MK, Lee JM, Lee JY. A phase II study of induction PD-1 blockade (nivolumab) in patients with surgically completely resectable mismatch repair deficient endometrial cancer (NIVEC). J Gynecol Oncol. 2025 May;36(3):e35. doi: 10.3802/jgo.2025.36.e35. Epub 2024 Oct 23. PMID 39530558